CLINICAL TRIAL: NCT03366987
Title: Nonalcoholic Fatty Liver Disease is Associated With Increased Atrial Fibrillation Risk in an Elderly Chinese Population: a Cross-sectional Study
Brief Title: Nonalcoholic Fatty Liver Disease is Associated With Increased Atrial Fibrillation Risk in an Elderly Chinese Population
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ningbo2
Record Dates: First submitted 2017-10-26; First posted 2017-12-08 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2018-07

CONDITIONS: Nonalcoholic Fatty Liver Disease; Atrial Fibrillation; Cross-sectional Study
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Atrial fibrillation and nonalcoholic fatty liver disease are two pathological conditions that are highly prevalent worldwide and share multiple CVD risk factors. There is rare research performed among elderly adults. The investigators are conducting a cross-sectional analysis of elderly adults (≥65 years) to investigate the association between atrial fibrillation and nonalcoholic fatty liver disease in an elderly Chinese population.

DETAILED DESCRIPTION:
Because of the aging population and improvements in cardiovascular treatments, its prevalence is expected to increase substantially over the next few decades. AF has been reported to be associated with high rates of hospitalization and death. Along with older age, there are many independent risk factors for AF like obesity, hypertension, diabetes, ischemic heart disease, heart failure and valvular heart disease.

Non-alcoholic fatty liver disease is one of the most prevalent liver diseases in the world whose prevalence ranges from 6% to 35%, with a median of 20% in the general population. In recent years, an increasing body of evidence have indicated that NAFLD is linked to cardiovascular disease, myocardial abnormalities, left ventricular diastolic dysfunction, heart failure, aortic valve sclerosis and so on.

NAFLD has also been observed to be significantly associated with AF in patients with type 2 diabetes. Furthermore, a cohort study showed that NAFLD was associated with an increased risk of prevalent AF in a middle-aged population. However, whether the association between NAFLD and AF also holds true in the elderly population remains uncertain. Therefore, the investigators conducted this cross-sectional study to explore the association between NAFLD and AF in an elderly Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* those who undergone an annual physical examination at Zhenhai Lianhua Hospital, Ningbo, China in 2014
* elderly adults (≥65 years old)

Exclusion Criteria:

* unknown alcohol intake or excessive alcohol intake
* unknown BMI or BMI≤18.0kg/m2
* incomplete basic physical data
* missing liver ultrasonic diagnosis
* unknown causes of chronic liver disease

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The elderly adults (≥65 years old) who had undergone an annual physical examination at Zhenhai Lianhua Hospital, Ningbo, China in 2014
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Association of nonalcoholic fatty liver disease and atrial fibrillation | the physical examination data in the year of 2014
  The association of nonalcoholic fatty liver disease and atrial fibrillation by chi-square test.

SECONDARY OUTCOMES:
Prevalence of AF in an elderly Chinese population stratified by normal or elevated serum liver enzyme concentration | the physical examination data in the year of 2014
  Prevalence of AF in an elderly Chinese population stratified by normal or elevated serum liver enzyme concentration by chi-square test.
Prevalence of AF in an elderly Chinese population stratified by NAFLD status on ultrasound combined with normal or elevated serum AST/ALT/GGT concentration | the physical examination data in the year of 2014
  Prevalence of AF in an elderly Chinese population stratified by NAFLD status on ultrasound combined with normal or elevated serum AST/ALT/GGT concentration by chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xu, Dr., Principal Investigator — Department of Gastroenterology, Ningbo No. 1 Hospital, Ningbo, China
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol (2017-12-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03366987/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03366987/SAP_001.pdf